CLINICAL TRIAL: NCT04793022
Title: A Prospective Clinical Trial Comparing General Anesthesia With Interscalene Nerve Block vs. Deep Sedation Via TIVA-P With Interscalene Nerve Block in Outpatient Shoulder Arthroscopies
Brief Title: Total Intravenous Anesthesia With Propofol vs. General Anesthesia in Outpatient Shoulder Arthroscopic Surgeries
Acronym: TIVA
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Carilion Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB19-471
Record Dates: First submitted 2021-02-22; First posted 2021-03-11 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-01

CONDITIONS: Rotator Cuff Tears; Rotator Cuff Injuries; Orthopedic Disorder; Sports Injury; Anesthesia
MeSH Terms: conditions — Rotator Cuff Injuries; Musculoskeletal Diseases; Athletic Injuries | interventions — Propofol; Anesthesia, General

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- TIVA-Propofol (Experimental): Intravenous anesthesia with Propofol
  Interventions: Drug: TIVA with Propofol
- Inhaled Anesthesia (Active Comparator): General Inhaled Anesthesia
  Interventions: Drug: Inhaled Anesthesia

INTERVENTIONS:
Drug: TIVA with Propofol — Total intravenous anesthesia with propofol
  Other Names: Propofol
  Arms: TIVA-Propofol
Drug: Inhaled Anesthesia — General anesthesia given with inhaled anesthetics
  Other Names: General Anesthesia
  Arms: Inhaled Anesthesia

SUMMARY:
This study is comparing total intravenous anesthesia with propofol with a regional nerve block against general anesthesia with a regional nerve block on the primary endpoint of time to meet discharge criteria.

DETAILED DESCRIPTION:
The primary objective of this study is to determine if using Total Intravenous Anesthesia with Propofol (TIVA-P sedation) with a regional nerve block will decrease the time to meet discharge criteria. This will be done with patients undergoing shoulder arthroscopic procedures at the Roanoke Ambulatory Surgical Center. Currently, inhaled general anesthesia (GA) with a regional nerve block is utilized for these outpatient arthroscopic procedures. This involves the patient receiving Propofol through an IV to put a patient to sleep, followed by intubation (breathing tube in throat) and the administration of inhaled anesthesia for the duration of the procedure. Another approach for anesthesia in these procedures is TIVA-P sedation. In this protocol the patient receives the same initial amount of Propofol through the IV as they would if they were getting general anesthesia. Once they are asleep, it is maintained with a continuous intravenous administration of Propofol. With this approach, the patient is not intubated and exposed to the same anesthetic agents as general anesthesia. As a result, the patient may not experience the potential side effects associated with general anesthesia. We believe that this will lead to a faster time to meet discharge criteria and also fewer of anesthetic side effects.

ELIGIBILITY:
Inclusion Criteria:

* 18-75 years of age
* Candidate for a shoulder arthroscopic procedure in the beach chair position

Exclusion Criteria:

* American Society of Anesthesiologists (ASA) level 4 or above
* History of brachial plexus injury
* Chronic Obstructive Pulmonary Disorder
* Unstable Asthma
* BMI greater than 40
* Allergy to local anesthesic (bupivacaine)
* Contralateral phrenic nerve impairment
* History of Difficult Airway
* Poorly Controlled Gastroesophageal Reflux Disease
* Known Aspiration Risk
* Surgery not performed at the Roanoke Ambulatory Surgical Center
* Pregnant patients or patients who have a positive pre-operative human chorionic gonadotropin (beta-HCG) pregnancy test
* Coagulopathies
* Allergy to propofol
* Patient request for specific anesthesia method

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 192 (Estimated)
Dates: Start 2021-02-02 (Actual); Primary Completion 2023-08-01 (Estimated); Study Completion 2023-08-01 (Estimated)

PRIMARY OUTCOMES:
Time to meet discharge criteria | Immediately after the intervention/procedure/surgery
  How long it takes until the patient is ready to be discharged from the PACU

SECONDARY OUTCOMES:
Pain Scale | Baseline, pre-intervention/procedure/surgery, and up to 21 days after procedure.
  Pain measured via pain scale: 0 through 5. 0 is no pain, 5 is worst pain ever felt.
Number of procedures requiring anesthetic intervention during surgery | During the intervention/procedure/surgery
  Use of preoperative interventions including vasopressors, antiemetics, sedatives
Satisfaction scale | Up to 21 days after procedure.
  How satisfied the patient is with their treatment, scale is rated "1-Poor, 2-Average, 3-Good, 4-Excellent" with higher numbers equating to more patient satisfaction.
post-anaesthesia care unit (PACU) I to post-anaesthesia care unit (PACU) II transition time | Immediately after the intervention/procedure/surgery
  The amount of time it takes to go from PACU I to PACU II
Antiemetic use in PACU | Immediately after the intervention/procedure/surgery
  Counting dosage of antiemetic use in PACU.
Surgical time | During the intervention/procedure/surgery
  Time patient is in surgery.

CONTACTS AND LOCATIONS:
Overall Officials: John Tuttle, MD, MS, Principal Investigator — Carilion Clinic Ortho Surgeon
Locations (1):
- Carilion Clinic Institute of Orthopedics and Neurosurgery, Roanoke, Virginia, United States

IPD SHARING:
Plan to Share IPD: No
Data will be collected, de-identified, and published in a manuscript once the study is completed.